CLINICAL TRIAL: NCT01642589
Title: Safety and Immunogenicity Study for Use of Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) Versus Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Adacel®) in Subjects 11 to 55 Years of Age in South Korea
Brief Title: Safety and Immunogenicity Study for Use of Menactra® Versus Adacel® in Subjects 11 to 55 Years of Age in South Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTA52; U1111-1122-2028 (Other: WHO)
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Meningitis; Meningococcal Disease
Keywords: Meningitis; Meningococcal disease; Menactra®; Adacel®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines; Tetanus Toxoid; adacel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menactra® Group (Experimental): Participants will receive Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®)
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®)
- Tdap - Adacel® Group (Active Comparator): Participants will receive Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Tdap - Adacel®)
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed — 0.5 mL, Intramuscular
  Other Names: Adacel®
  Arms: Tdap - Adacel® Group

SUMMARY:
The aim of the study is to assess safety and immunogenicity of a single dose of Menactra® in support of registration of the vaccine in South Korea.

Primary Objective:

* To demonstrate that the seroconversion rate is higher than 60% for serogroups A, C, Y and W-135, 28 days after a single dose of Menactra®.

Secondary objectives:

* To demonstrate the superiority of Menactra® versus Adacel® in terms of seroconversion rate for serogroups A, C, Y, and W-135, 28 days after a single dose of vaccine
* To describe the safety profile after 1 dose of Menactra® or Adacel® vaccine.
* To describe the Serum Bactericidal Assay Using Baby Rabbit (SBA-BR) Complement titers before and 28 days after a single dose of Menactra® or Adacel® vaccine.

DETAILED DESCRIPTION:
All participants will receive a single dose of vaccine, and will be assessed for immunogenicity at baseline (pre-vaccination) and at 28 days post-vaccination.

Safety data, including serious adverse events (SAEs) will be collected for Day 0 through Day 28 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11 to 55 years on the day of inclusion
* Subject aged 11 to 19 years: assent form signed and dated by the subject and informed consent form signed and dated by at least 1 parent or another legal representative
* Subject aged 20 to 55 years: informed consent form signed and dated by the subject

If the subject or the subject's parent(s) or legal representative is illiterate, an independent witness is required to sign the consent form.

* Subject and parent/legally acceptable representative (if applicable) are able to attend all scheduled visits and comply with all trial procedures
* Covered by health insurance.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of child-bearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post menopausal for at least 1 year, surgically sterile (hysterectomy or bilateral tubal ligation), or using an effective method of contraception or abstinence for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination)
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure
* Receipt or planned receipt of any vaccine in the 4 weeks preceding or following the trial vaccination. Monovalent pandemic influenza vaccines and multivalent pandemic influenza vaccines can be administered at any time during the study
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine
* Vaccination against diphtheria or tetanus in the past 5 years or any previous vaccination with either Adacel® or any other Tdap vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of invasive meningococcal disease, confirmed either clinically, serologically, or microbiologically
* At high risk for invasive meningococcal disease during the trial
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia, bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Received oral or injectable antibiotic therapy within the 72 hours prior to the first blood draw
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Personal history of Guillain-Barré Syndrome.

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (7):
- South Korea (7):
  - Incheon, Chung gu
  - Gyeonggi-do, Dongan Gu Anyang
  - Seoul, Dongdaemun gu
  - Seoul, Seodaemun gu
  - Seoul, Seongbuk gu
  - Gyeonggi-do, Suwon
  - Gangwon Do, Wonju

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 13 July 2012 to 17 December 2012 in 8 clinic centers in South Korea.
Pre-assignment Details: A total of 300 participants that met all inclusion but none of the exclusion criteria were randomized and vaccinated in this study
Groups:
- Menactra® Group: Participants received Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®)
- Tdap - Adacel® Group: Participants received Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Tdap - Adacel®)
Period: Overall Study
Arm/Group | Menactra® Group | Tdap - Adacel® Group
Started | 200 | 100
Completed | 199 | 99
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Group | Tdap - Adacel® Group | Total
Number analyzed (Participants) | 200 | 100 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 49 | 149
  Between 18 and 65 years | 100 | 51 | 151
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 24.9 (11.5) | 24.2 (10.1) | 24.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 58 | 165
  Male | 93 | 42 | 135
Region of Enrollment [Number; unit: Participants]
  Korea, Republic of | 200 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion Following Vaccination With Either Menactra® or Adacel® Vaccine
Description: Functional antibody activity for anti-meningococcal antibody to serogroups A, C, Y, and W-135 were measured using the Serum bactericidal assay using baby rabbit complement (SBA-BR).
  Seroconversion was defined as post-vaccination antibody titers of ≥ 4-fold increase from pre-vaccination level.
Time Frame: 28 Days post-vaccination
Population: Functional antibody activity for anti meningococcal antibody to serogroups A, C, Y, and W 135 were determined in the Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Menactra® Group | Tdap - Adacel® Group
Number analyzed (Participants) | 200 | 100
Percentage of participants
  Serogroup A | 78 | 9 [0 to 0]
  Serogroup C | 88 | 8 [0 to 0]
  Serogroup Y | 75 | 12 [0 to 0]
  Serogroup W-135 | 92 | 8 [0 to 0]

2. Secondary Outcome: Percentage of Participants With Functional Antibody Titers at ≥1:8 Dilution Before and After Menactra® or Adacel® Vaccination
Description: Functional antibody activity for anti-meningococcal antibody to serogroups A, C, Y, and W-135 were measured using the Serum bactericidal assay using baby rabbit complement (SBA-BR) at ≥ 1:8 dilution.
Time Frame: Day 0 (pre-vaccination) and 28 days post-vaccination
Population: Functional antibody activity for anti-meningococcal antibody to serogroups A, C, Y, and W-135 were determined in the Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Menactra® Group | Tdap - Adacel® Group
Number analyzed (Participants) | 200 | 100
Percentage of participants
  Serogroup A (Pre-vaccination) | 68 | 76 [0 to 0]
  Serogroup A (Post-vaccination) | 100 | 78 [0 to 0]
  Serogroup C (Pre-vaccination) | 28 | 19 [0 to 0]
  Serogroup C (Post-vaccination) | 93 | 24 [0 to 0]
  Serogroup Y (Pre vaccination) | 75 | 75 [0 to 0]
  Serogroup Y (Post-vaccination) | 99 | 81 [0 to 0]
  Serogroup W-135 (Pre-vaccination) | 50 | 44 [0 to 0]
  Serogroup W-135 (Post-vaccination) | 98 | 48 [0 to 0]

3. Secondary Outcome: Percentage of Participants With Functional Antibody Titers at ≥1:128 Dilution Before and After Menactra® or Adacel® Vaccination.
Description: Functional antibody activity for anti-meningococcal antibody to serogroups A, C, Y, and W-135 were measured using the Serum bactericidal assay using baby rabbit complement (SBA-BR) at ≥ 1:128 dilution.
Time Frame: Day 0 (pre-vaccination) and 28 days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Menactra® Group | Tdap - Adacel® Group
Number analyzed (Participants) | 200 | 100
Percentage of participants
  Serogroup A (Pre-vaccination) | 57 | 64 [0 to 0]
  Serogroup A (Post-vaccination) | 99 | 70 [0 to 0]
  Serogroup C (Pre-vaccination) | 25 | 15 [0 to 0]
  Serogroup C (Post-vaccination) | 89 | 16 [0 to 0]
  Serogroup Y (Pre-vaccination) | 52 | 48 [0 to 0]
  Serogroup Y (Post-vaccination) | 96 | 57 [0 to 0]
  Serogroup W 135 (Pre-vaccination) | 22 | 25 [0 to 0]
  Serogroup W 135 (Post-vaccination) | 95 | 27 [0 to 0]

4. Secondary Outcome: Geometric Mean Titers of Serum Bactericidal Assay Using Baby Rabbit Complement (SBA-BR) Antibody Against Serogroups A, C, Y, and W-135 Before and After Menactra® or Adacel® Vaccination
Description: Functional antibody activity for anti-meningococcal antibody to serogroups A, C, Y, and W-135 were measured using the Serum bactericidal assay using baby rabbit complement (SBA-BR).
Time Frame: Day 0 (pre-vaccination) and 28 days post-vaccination
Population: Geometric mean titers for the anti meningococcal antibody to serogroups A, C, Y, and W 135 were determined in the Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra® Group | Tdap - Adacel® Group
Number analyzed (Participants) | 200 | 100
Titers
  Serogroup A (pre-vaccination) | 46.1 [33.7 to 63.2] | 75.6 [48.9 to 117]
  Serogroup A (post-vaccination) | 1121 [949 to 1324] | 87.6 [57.1 to 135]
  Serogroup C (pre-vaccination) | 5.80 [4.50 to 7.46] | 4.63 [3.26 to 6.56]
  Serogroup C (post-vaccination) | 667 [504 to 884] | 5.64 [3.82 to 8.32]
  Serogroup Y (pre-vaccination) | 50.1 [37.7 to 66.6] | 47.2 [31.9 to 69.8]
  Serogroup Y (post-vaccination) | 620 [521 to 738] | 66.8 [45.5 to 98.0]
  Serogroup W-135 (pre-vaccination) | 13.0 [9.83 to 17.1] | 11.9 [7.79 to 18.1]
  Serogroup W-135 (post-vaccination) | 851 [690 to 1050] | 14.9 [9.50 to 23.4]

5. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Events Following Vaccination With Either Menactra® or Adacel® Vaccine
Description: Solicited injection site reactions: Pain, Redness, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia.
  Grade 3 injection site reactions: Pain - Significant, prevents daily activity; Redness and Swelling - > 100 mm. Grade 3 Systemic reactions: Fever - ≥ 39.0°C; Headache, Malaise, and Myalgia - Significant, prevents daily activity.
Time Frame: Day 0 up to Day 28 post-vaccination
Population: Solicited injection site and systemic events were assessed in all randomized and vaccinated study participants, Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Menactra® Group | Tdap - Adacel® Group
Number analyzed (Participants) | 200 | 100
Participants
  Injection Site Pain (199, 99) | 64 | 72 [0 to 0]
  Grade 3 Injection Site Pain (199, 99) | 1 | 2 [0 to 0]
  Injection Site Erythema (199, 99) | 5 | 9 [0 to 0]
  Grade 3 Injection Site Erythema (199, 99) | 0 | 0 [0 to 0]
  Injection Site Swelling (199, 99) | 3 | 6 [0 to 0]
  Grade 3 Injection Site Swelling (199, 99) | 0 | 0 [0 to 0]
  Fever (199, 99) | 0 | 3 [0 to 0]
  Grade 3 Fever (199, 99) | 0 | 0 [0 to 0]
  Headache (199, 99) | 37 | 24 [0 to 0]
  Grade 3 Headache (199, 99) | 2 | 1 [0 to 0]
  Malaise (199, 99) | 36 | 23 [0 to 0]
  Grade 3 Malaise (199, 99) | 1 | 1 [0 to 0]
  Myalgia (199, 99) | 51 | 42 [0 to 0]
  Grade 3 Myalgia (199, 99) | 1 | 1 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination
Arm/Group | Menactra® Group | Tdap - Adacel® Group
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/100
Other Adverse Events (participants affected / at risk) | 92/200 | 76/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Menactra® Group (N=200) | Tdap - Adacel® Group (N=100)
Injection Site Pain (General disorders) | 64/199 (64) | 72/99 (72)
Injection Site Erythema (General disorders) | 5/199 (5) | 9/99 (9)
Injection Site Swelling (General disorders) | 3/199 (3) | 6/99 (6)
Headache (Nervous system disorders) | 37/199 (37) | 24/99 (24)
Malaise (General disorders) | 36/199 (36) | 23/99 (23)
Myalgia (Musculoskeletal and connective tissue disorders) | 51/199 (51) | 42/99 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.